CLINICAL TRIAL: NCT01145222
Title: A Phase IIb Study Evaluating the Safety and Efficacy of Multiple Doses of CNS 7056 Compared to Midazolam in Patients Undergoing Colonoscopy
Brief Title: Multiple Dose Safety and Efficacy Study Evaluating CNS 7056 Versus Midazolam in Patients Undergoing Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNS 7056-004
Record Dates: First submitted 2010-05-27; First posted 2010-06-16 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Sedation
Keywords: CNS 7056; Procedural Sedation; Colonoscopy
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A. Remimazolam (CNS 7056) (Experimental): Initial 8 mg iv for sedation induction, and 3 mg iv top-ups for sedation maintenance.
  Fentanyl pre-treatment: up to 100 μg (at the discretion of the investigator) and 25 μg top-up doses.
  Interventions: Drug: A. CNS 7056
- B. Remimazolam (CNS 7056) (Experimental): Initial 7 mg iv for sedation induction, and 2 mg iv top-ups for sedation maintenance.
  Fentanyl pre-treatment: up to 100 μg (at the discretion of the investigator) and 25 μg top-up doses.
  Interventions: Drug: B. CNS 7056
- C. Remimazolam (CNS 7056) (Experimental): Initial 5 mg iv for sedation induction, and 3 mg iv top-ups for sedation maintenance.
  Fentanyl pre-treatment: up to 100 μg (at the discretion of the investigator) and 25 μg top-up doses.
  Interventions: Drug: C. CNS 7056
- D. Midazolam (Active Comparator): Initial 2.5 mg iv for sedation induction, and 1 mg iv top-ups for sedation maintenance.
  Fentanyl pre-treatment: up to 100 μg (at the discretion of the investigator) and 25 μg top-up doses
  Interventions: Drug: D. Midazolam

INTERVENTIONS:
Drug: A. CNS 7056 — Initial low dose plus supplemental doses as necessary.
  Other Names: CAS No. 1001415-66-2; Remimazolam
  Arms: A. Remimazolam (CNS 7056)
Drug: B. CNS 7056 — Initial intermediate dose plus supplemental doses as necessary.
  Other Names: CAS No. 1001415-66-2; Remimazolam
  Arms: B. Remimazolam (CNS 7056)
Drug: C. CNS 7056 — Initial high dose plus supplemental doses as necessary.
  Other Names: CAS No. 1001415-66-2; Remimazolam
  Arms: C. Remimazolam (CNS 7056)
Drug: D. Midazolam — Initial standardized dose plus supplemental doses as necessary.
  Other Names: CAS No. 59467-96-8
  Arms: D. Midazolam

SUMMARY:
The purpose of this dose-response study is to assess the safety and efficacy of CNS 7056 compared with midazolam to maintain suitable sedation levels in patients undergoing colonoscopy.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel group, dose-response study to assess the safety and efficacy of three dose levels of CNS 7056 compared with midazolam to maintain suitable sedation levels in patients undergoing colonoscopy.

Safety assessment will include physical examinations, vital signs, ECGs, pulse oximetry measurements, capnography, clinical chemistry and hematology laboratory tests, routine drug and ethanol screening, urinalysis, pregnancy test, pain on injection using a verbal scale, and monitoring of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 18 to 70 years inclusive, scheduled to undergo a standard colonoscopy.
* American Society of Anesthesiologists Physical Status (ASA PS) Score I, II, or III.
* Weight range 55 to 130 kg inclusive.
* Body mass index (BMI) range 18 to 33 kg/m2 inclusive
* Patients of child-bearing potential and their partners must have been willing to use adequate contraception such as an intrauterine device, diaphragm or condom during the study and until 1 month after the last study drug administration. Childbearing potential was defined as "all patients unless they were a female post menopausal for at least 2 years, or were surgically sterile."
* Patient voluntarily signed and dated an ICF that was approved by an IRB prior to the conduct of any study procedure.
* Patient was willing and able to comply with study requirements and return for a Follow up Visit (Day 4 ± 3 day) after the colonoscopy.

Exclusion Criteria:

* Expected duration of colonoscopy > 30 minutes.
* Patients with a suspected or diagnosed pathology of the lower GI tract that would have added to the risk of colonoscopy, such as strictures, active inflammatory bowel disease.
* ASA III patients with history of sleep apnea.
* ASA III patients with obesity (BMI ≥ 30 kg/m2).
* Patients with evidence of uncontrolled renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction, or other clinically significant (CS) findings at screening that, in the investigator's or medical monitor's opinion, should have excluded them from the study.
* Patients with clinically significant abnormalities in 12 lead ECG recorded at screening.
* Female patients with a positive serum human chorionic gonadotropin (HCG) pregnancy test at screening or baseline.
* Lactating female patients.
* Patients with positive drugs of abuse screen at baseline.
* Patients with positive serum ethanol at baseline.
* Patient with a history of drug or ethanol abuse.
* Patients in receipt of any investigational drug within 30 days or less than 7 half lives (whichever was longer) before the start of the study, or scheduled to receive one during the study period.
* Patients with a known sensitivity to benzodiazepines, flumazenil, opioids, naloxone, or a medical condition such that these agents were contraindicated.
* Patients with an inability to communicate well with the investigator.
* Patients in whom management of airway was judged to be difficult due to, e.g., thyro-mental distance ≤ 4 cm ("short neck"), or Mallampati score of 4.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Helen Keller Hospital, Sheffield, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - ACRI Phase I LLC, Anaheim, California
  - Advanced Clinical Research Associates, Anaheim, California
  - Miami Research Associates, South Miami, Florida
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Options Health Research, Tulsa, Oklahoma
  - Charlottesville Medical Research, Charlottesville, Virginia

REFERENCES:
- [Result] Pambianco DJ, Borkett KM, Riff DS, Winkle PJ, Schwartz HI, Melson TI, Wilhelm-Ogunbiyi K. A phase IIb study comparing the safety and efficacy of remimazolam and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2016 May;83(5):984-92. doi: 10.1016/j.gie.2015.08.062. Epub 2015 Sep 9. PMID 26363333

RESULTS

PARTICIPANT FLOW:
Groups:
- Remimazolam 8.0/3.0 mg: Double-blind Remimazolam iv arm: 8 mg for sedation induction, and 3 mg top-ups for sedation maintenance
- Remimazolam 7.0/2.0 mg: Double-blind Remimazolam iv arm: 7 mg for sedation induction, and 2 mg top-ups for sedation maintenance
- Remimazolam 5.0/3.0 mg: Double-blind Remimazolam iv arm: 5 mg for sedation induction, and 3 mg top-ups for sedation maintenance
- Midazolam 2.5/1.0: Double-blind Midazolam iv arm: 2.5 mg for sedation induction, and 1.0 mg top-ups for sedation maintenance.
Period: Overall Study
Arm/Group | Remimazolam 8.0/3.0 mg | Remimazolam 7.0/2.0 mg | Remimazolam 5.0/3.0 mg | Midazolam 2.5/1.0
Started | 40 | 40 | 41 | 41
Safety Population (Safety population included all randomized patients who received any amount of study drug) | 40 | 40 | 40 | 41
Intention to Treat (ITT) Population (Received any amount of study drug, started the procedure, and had at least 1 efficacy assessment) | 40 | 40 | 40 | 40
Completed | 40 | 40 | 40 | 40
Not Completed | 0 | 0 | 1 | 1
Not completed — Procedure not done (no anesthesiologist) | 0 | 0 | 1 | 0
Not completed — Poor bowel preparation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is the Safety Population
Groups:
- Midazolam 2.5/1.0: Double-blind Midazolam iv arm: 2.5 mg for sedation induction, and 1 mg top-ups for sedation maintenance.
- Total: Total of all reporting groups
Arm/Group | Remimazolam 8.0/3.0 mg | Remimazolam 7.0/2.0 mg | Remimazolam 5.0/3.0 mg | Midazolam 2.5/1.0 | Total
Number analyzed (Participants) | 40 | 40 | 40 | 41 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.22) | 54.5 (8.07) | 54.0 (10.30) | 55.5 (5.86) | 54.6 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 22 | 20 | 89
  Male | 18 | 15 | 18 | 21 | 72
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 41 | 161
Height [Mean (Standard Deviation); unit: cm] | 169.15 (11.0) | 168.18 (8.3) | 169.01 (11.3) | 169.87 (10.1) | 169.06 (10.2)
Weight [Mean (Standard Deviation); unit: kg] | 79.68 (13.4) | 76.23 (11.6) | 76.79 (14.5) | 76.95 (13.6) | 77.41 (13.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 27.79 (3.451) | 27.02 (4.042) | 26.73 (3.063) | 26.58 (3.515) | 27.03 (3.533)

OUTCOME MEASURES:

1. Primary Outcome: Success Rates of the Procedure
Description: Success of the procedure is a composite endpoint consisting of: Modified Observer's Assessment for Alertness/Sedation (MOAA/S) scores ≤4 on three consecutive measurements after administration of study drug AND completion of the endoscopy procedure AND no requirement for rescue sedative medication AND no requirement for manual or mechanical ventilation
Time Frame: From start of study drug injection to patient discharge
Population: Analysis Population is the ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Remimazolam 8.0/3.0 mg | Remimazolam 7.0/2.0 mg | Remimazolam 5.0/3.0 mg | Midazolam 2.5/1.0
Number analyzed (Participants) | 40 | 40 | 40 | 40
Participants | 37 | 38 | 39 | 30
Statistical Analysis 1: Comparison: Remimazolam 8.0/3.0 mg vs Remimazolam 7.0/2.0 mg vs Remimazolam 5.0/3.0 mg vs Midazolam 2.5/1.0; Test type: Superiority — Overall comparison between remimazolam and midazolam; p = 0.007, Fisher Exact

2. Secondary Outcome: Time to Fully Alert
Description: Time to first of 3 consecutive MOAA/S scores of 5 after the last injection of double-blind study medication
Time Frame: From last injection of double-blind study medication until fully alert criteria are reached
Population: Analysis Population is the ITT Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Remimazolam 8.0/3.0 mg | Remimazolam 7.0/2.0 mg | Remimazolam 5.0/3.0 mg | Midazolam 2.5/1.0
Number analyzed (Participants) | 40 | 40 | 40 | 40
minutes | 13.6 (7.48) | 11.3 (5.69) | 13.3 (7.21) | 15.2 (7.43)

3. Secondary Outcome: Time to Ready for Discharge
Description: Time of the first of 3 consecutive Aldrete scores ≥ 9
Time Frame: After the Last Injection of Double-Blind Study Medication AND after end of colonoscopy until first of 3 consecutive Aldrete scores ≥ 9
Population: Analysis Population is the ITT Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Remimazolam 8.0/3.0 mg | Remimazolam 7.0/2.0 mg | Remimazolam 5.0/3.0 mg | Midazolam 2.5/1.0
Number analyzed (Participants) | 40 | 40 | 40 | 40
minutes
  After last injection | 14.6 (8.52) | 12.4 (6.72) | 11.3 (4.86) | 15.3 (8.13)
  After end of colonoscopy | 5.0 (6.29) | 4.6 (4.58) | 3.8 (4.16) | 5.5 (6.59)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) were collected from first dose of study drug until Day 4 ± 3 days, and were followed until resolution of any ongoing TEAE up to 30 days
Description: Total number of participants affected with Other (Not Including Serious) Adverse Events represents overall number of participants with non-serious TEAEs reported with a threshold of 5% in any of the arms
Arm/Group | Remimazolam 8.0/3.0 mg | Remimazolam 7.0/2.0 mg | Remimazolam 5.0/3.0 mg | Midazolam 2.5/1.0
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 10/40 | 8/40 | 9/40 | 6/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remimazolam 8.0/3.0 mg (N=40) | Remimazolam 7.0/2.0 mg (N=40) | Remimazolam 5.0/3.0 mg (N=40) | Midazolam 2.5/1.0 (N=41)
Bradycardia (Cardiac disorders) | 3 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 2
Headache (Nervous system disorders) | 1 | 3 | 3 | 2
Hypertension (Vascular disorders) | 3 | 0 | 1 | 4
Nausea (Gastrointestinal disorders) | 3 | 2 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submission for publication, presentation or use, sponsor shall review and comment any proposed oral or written publication, which period may be extended for an additional 30 days. To seek patent protection, sponsor shall have the right to delay the proposed publication for an additional 60 days.